CLINICAL TRIAL: NCT03190356
Title: Soberlink - MAP Outcomes Study Protocol
Status: Terminated | Type: Observational
Why Stopped: Business Decision
Sponsor: Soberlink Healthcare LLC (Industry)
Collaborators: MAP Health Management LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: SLMAPPROT-2017-001
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Alcohol Addiction
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Primary diagnosis alcohol use disorder (AUD): Primary diagnosis of alcohol use disorder (AUD) population enrolled in MAP's System
  Interventions: Device: Soberlink Cellular Device
- Secondary diagnosis alcohol use disorder (AUD): Secondary diagnosis of alcohol use disorder (AUD) population enrolled in MAP's System
  Interventions: Device: Soberlink Cellular Device

INTERVENTIONS:
Device: Soberlink Cellular Device — Soberlink Cellular Device delivers real-time blood alcohol results to people who support individuals in recovery. MAP platform helps monitor and support compliance with discharge plans while providing tools to improve outcomes for behavioral health diagnoses.
  Other Names: MAP patient engagement platform (EHR)

SUMMARY:
The purpose of this study is to show the effectiveness of Soberlink's remote alcohol monitoring system integrated with MAP's patient engagement platform (EHR) to monitor a sample size of at-risk alcohol use disorder (AUD) population. Ultimately, this data is leveraged to improve clinical outcomes and manage financial risk through facilitating early interventions and other means of mitigating recidivism and costly treatment episodes from AUD population.

DETAILED DESCRIPTION:
The study will include 30 Clients with a primary or secondary diagnosis of alcohol use disorder (AUD) and are enrolled in MAP's System where dedicated Case Managers are monitoring the Client's relapse risk levels. Soberlink's remote alcohol system will provide data to inform the Case Manager if the Client has relapsed or is at risk of relapsing through the use of testing data compiled by the Soberlink System. Integrating Soberlink results into MAP's EMR will allow Case Manager to make better clinical decisions and reduce costs by mitigating the chances recidivism through early intervention. Clients will use the Soberlink Device for a period of 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between ages of 21-65 years old
* Subject is active in MAP's program with recovery support services
* Subject has received acute professional treatment in the last 120 days
* Primary or secondary diagnosis is Alcohol Use Disorder
* Subject willing to use Soberlink Device to provide BAC
* Subject is willing to discuss Soberlink test results with case manager
* Subject is willing to sign a Soberlink Client Agreement
* Subject is English speaking and reading

Exclusion Criteria:

* Alcohol Use Disorder is not a primary or secondary diagnosis
* Subject is currently taking anti-alcohol medications
* Subject will not be in the United States through duration of study
* Subject is unwilling to properly use the device
* Subject is non-English speaking and reading
* Subject is a child, adolescent, cognitively impaired, diagnosed with a mental disorder, such as schizophrenia

Ages: 21 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 adult male/female clients with a primary or secondary diagnosis of alcohol use disorder (AUD) and are enrolled in MAP's System where dedicated Case Managers are monitoring the Client's relapse risk levels.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Recidivism | 90 days duration of subject participation
  Determination of client relapse or risk of relapsing through the use of testing data compiled by the Soberlink Cellular Device

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Hanrahan, PhD, Principal Investigator — Shannon Hanrahan
Locations (1):
- MAP Health Management LLC, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: American Cancer Society - Alcohol Use and Cancer — https://www.cancer.org/cancer/cancer-causes/diet-physical-activity/alcohol-use-and-cancer.html